CLINICAL TRIAL: NCT06397573
Title: Phase 1 Trial of Ablative Stereotactic MR-Guided Adaptive Reirradiation for Abdominal and Pelvic Tumors
Brief Title: Ablative Stereotactic MR-Guided Adaptive Reirradiation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Baptist Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-CHU-001
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Abdominal Cancer; Pelvic Cancer
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Re-Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablative Reirradiation (Experimental)
  Interventions: Radiation: Reirradiation

INTERVENTIONS:
Radiation: Reirradiation — Ablative reirradiation of 50 Gy in 5 fractions (5 sessions) that will occur once per day, either for 5 days in a row, or every other day.

SUMMARY:
This research study will enroll people who have cancer in their abdomen or pelvis that was treated previously with radiation therapy. The purpose of this research study is to test the safety and possible harms of treating tumors in these regions with another round of radiation therapy, called reirradiation or "reRT." The researchers want to find out what effects (good and bad) reRT has in people with cancer in the abdomen and pelvis.

ELIGIBILITY:
Inclusion Criteria:

* A primary or metastatic lesion in the abdomen or pelvis for which reirradiation will be delivered. There is no maximum lesion size.
* Single course of prior radiation therapy with prescribed equivalent dose in 2 Gy fractions (EDQ210) of at least 40 Gy.
* 50% isodose line of the prior radiation therapy course is expected to overlap at minimum the 50% isodose line of the radiation therapy delivered in this study.
* At least 6 months from completion of prior radiation therapy to initiation of study therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Life expectancy at least 6 months.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Abstinence is acceptable if it is the participant's preferred method. Should a participant become pregnant or suspect pregnancy while participating in this study, the treating physician must be informed immediately.
* Concurrent hormonal therapy or immunotherapy such as immune checkpoint inhibitor is allowed

Exclusion Criteria:

* Contraindication to having an MRI scan.
* Lesion that would receive study therapy arises from or invades a gastrointestinal (GI) luminal organ (a lesion abutting but not invading a GI luminal organ is permitted)
* Lesion that would receive study therapy is not located in the abdomen or pelvis.
* > 1 course of overlapping radiation therapy delivered to the abdomen or pelvis.
* < 70% of the gross tumor volume (GTV) receives at least the 95% of the prescribed dose on the original plan using the simulation day anatomy.
* More than 1 lesion in the abdomen or pelvis that requires reirradiation.
* History of inflammatory bowel disease.
* Unable to acquire DICOM radiation therapy treatment plan from the prior radiation therapy.
* Unresolved grade 2+ toxicity (Common Terminology Criteria for Adverse Events version 5.0) from previous anti-cancer therapy.
* Any condition in the opinion of the investigator that would interfere with evaluation of study treatment or interpretation of participant safety or study results.
* Individuals who are pregnant.
* Chemotherapy given within 1 week prior to or following reirradiation.
* Vascular endothelial growth factor (VEGF) inhibitor given within 8 weeks prior to or following reirradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or higher acute toxicity | 1 year
  Number of participants who experience Grade 3 or higher acute toxicity [graded per Common Terminology Criteria for Adverse Events (CTCAE)] possibly, probably, or definitely related to reRT.
Grade 5 toxicity | 1 year
  Number of participants who experience Grade 5 toxicity (graded per CTCAE) possibly, probably, or definitely related to reRT.

SECONDARY OUTCOMES:
Freedom from local progression (FFLP) | 1 year
  FFLP is defined as the duration of time from baseline to progressive disease (PD) in the re-irradiated lesion or death of any cause, whichever occurs first. Response to treatment will be assessed using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival (OS) | 1 year
  OS is defined as the defined as the duration of time from baseline to death of any cause, or date of last follow-up, whichever occurs first.
Grade 3 or higher late toxicity | 1 year
  Number of participants who experience Grade 3 or higher acute toxicity [graded per Common Terminology Criteria for Adverse Events (CTCAE)] possibly, probably, or definitely related to reRT that occurs at least 90 days after reRT therapy has ended.
Quality of life (QOL) | 1 year
  QOL will be assessed using the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire. The FACT-G is a 27-item questionnaire measuring physical, social, emotional, and functional well-being. All questions in the FACT-G use a 5-point rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a bit; and 4 = Very much), with a possible range of 0-108 points. Negatively worded items are reverse scored prior to summing so that higher scores indicate better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chuong, M.D., Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health South Florida, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt A, Das P, Minsky BD, Koay EJ, Krishnan S, Herman JM, Taniguchi C, Koong A, Smith GL, Holliday EB. Hyperfractionated abdominal reirradiation for gastrointestinal malignancies. Radiat Oncol. 2018 Aug 7;13(1):143. doi: 10.1186/s13014-018-1084-0. PMID 30086784
- [Background] Tao R, Tsai CJ, Jensen G, Eng C, Kopetz S, Overman MJ, Skibber JM, Rodriguez-Bigas M, Chang GJ, You YN, Bednarski BK, Minsky BD, Delclos ME, Koay E, Krishnan S, Crane CH, Das P. Hyperfractionated accelerated reirradiation for rectal cancer: An analysis of outcomes and toxicity. Radiother Oncol. 2017 Jan;122(1):146-151. doi: 10.1016/j.radonc.2016.12.015. Epub 2017 Jan 3. PMID 28057329
- [Background] Moningi S, Ludmir EB, Polamraju P, Williamson T, Melkun MM, Herman JD, Krishnan S, Koay EJ, Koong AC, Minsky BD, Smith GL, Taniguchi C, Das P, Holliday EB. Definitive hyperfractionated, accelerated proton reirradiation for patients with pelvic malignancies. Clin Transl Radiat Oncol. 2019 Aug 27;19:59-65. doi: 10.1016/j.ctro.2019.08.004. eCollection 2019 Nov. PMID 31517071
- [Background] Sadozye AH. Re-irradiation in Gynaecological Malignancies: A Review. Clin Oncol (R Coll Radiol). 2018 Feb;30(2):110-115. doi: 10.1016/j.clon.2017.11.013. Epub 2017 Dec 9. PMID 29233573
- [Background] Munoz F, Fiorica F, Caravatta L, Rosa C, Ferella L, Boldrini L, Fionda B, Alitto AR, Nardangeli A, Dionisi F, Arcangeli S, Di Marzo A, Pontoriero A, Donato V, Massaccesi M. Outcomes and toxicities of re-irradiation for prostate cancer: A systematic review on behalf of the Re-Irradiation Working Group of the Italian Association of Radiotherapy and Clinical Oncology (AIRO). Cancer Treat Rev. 2021 Apr;95:102176. doi: 10.1016/j.ctrv.2021.102176. Epub 2021 Mar 8. PMID 33743409
- [Background] Barsky AR, Reddy VK, Plastaras JP, Ben-Josef E, Metz JM, Wojcieszynski AP. Proton beam re-irradiation for gastrointestinal malignancies: a systematic review. J Gastrointest Oncol. 2020 Feb;11(1):187-202. doi: 10.21037/jgo.2019.09.03. PMID 32175122
- [Background] Abusaris H, Hoogeman M, Nuyttens JJ. Re-irradiation: outcome, cumulative dose and toxicity in patients retreated with stereotactic radiotherapy in the abdominal or pelvic region. Technol Cancer Res Treat. 2012 Dec;11(6):591-7. doi: 10.7785/tcrt.2012.500261. Epub 2012 May 7. PMID 22568625
- See also: Miami Cancer Institute — https://cancer.baptisthealth.net/miami-cancer-institute